CLINICAL TRIAL: NCT01813734
Title: A Phase II, Open-Label Study of Ponatinib, A Multi-Targeted Oral Tyrosine Kinase Inhibitor, in Advanced Non-Small Cell Lung Cancer Harboring RET Translocations
Brief Title: Ponatinib in Advanced NSCLC w/ RET Translocations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alice Shaw, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-103
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: RET gene mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ponatinib Treatment Arm (Experimental): Ponatinib 30 mg PO daily
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — 28 day cycle

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied.

It has been found that some people with NSCLC have a change (mutation) in a certain gene called the RET gene. This mutated gene may help cancer cells grow. Only participants with a RET mutation will be allowed to participate. In this study, investigators are testing the strategy of using a study drug designed to inhibit or shut off growth signals that results from the mutated RET gene.

Ponatinib is an anti-cancer drug that has been used in research studies for other types of cancer. Ponatinib blocks several growth signals in cancer cells, including RET. In this research study, investigators are looking to see whether ponatinib is effective and safe in treating NSCLC harboring RET rearrangements.

DETAILED DESCRIPTION:
Participants in this research study will be asked to undergo some screening tests or procedures to confirm that eligibility. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that participants do not take part in the research study. These tests and procedures include the following: medical history, vital signs, physical exam, performance status, electrocardiogram, echocardiogram, routine blood tests, pregnancy test and an assessment of tumor by CT or MRI. If these tests show that a participant is eligible to participate in the research study, he/she will begin the study treatment. If a patient does not meet the eligibility criteria, he/she will not be able to participate in this research study.

Participants will take the study drug once a day, every day of the cycle. Each treatment cycle lasts 28 days (4 weeks). Participants will be given a drug diary to record the drug they take each day. The diary will also include special instructions for taking the study drug.

For cycles 1-20, participants will visit the clinic to have tests and procedures done at the time points listed here: On Day 1-physical exam, vital signs, performance status, electrocardiogram, routine blood tests, pharmacokinetic test, clinical exam and assessment of tumor. On day 15 of cycle 1-vital signs, routine blood tests and clinical exam.

For cycles 11 and on, participants will visit the clinic every 6 weeks. Some of these visits will happen on Day 1 of the cycle and some of these visits will happen on Day 15 of the cycle. At each visit, the following tests and procedures will be done: physical exam, vital signs, performance status, electrocardiogram, routine blood tests, clinical exam, and an assessment of your tumor.

Participants will visit the clinic when their study doctor takes them off study drug permanently. They will also visit the clinic 30 days after stop taking the study drug. The following tests and procedures will be done: physical exam, vital signs, performance status, electrocardiogram, routine blood tests, pregnancy test, clinical exam and a tumor assessment.

Investigators would also like to keep track of participant's medical condition for two years after their first study dose. Investigators will contact participants by telephone every 3 months. If participants still come to the clinic, visits might be used as contact.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced NSCLC
* Molecular confirmation of a RET translocation
* At least one measurable lesion as defined by RECIST
* No restriction on number of prior therapies
* Estimated life expectancy of at least 12 weeks
* Able to swallow and retain orally administered medication
* Must agree to use an effective form of contraception from enrollment through 30 days after the end of study treatment
* Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities
* Pregnant or breastfeeding
* Major surgery within 28 days of initiating therapy
* History of CNS disease (Note: Participants with brain metastases will be eligible if treated appropriately and if they remain clinically stable).
* Anti-cancer therapy within 3 weeks
* History of significant bleeding disorder unrelated to cancer
* History of acute pancreatitis within 1 year of study entry or history of chronic pancreatitis
* History of alcohol abuse
* Uncontrolled hypertriglyceridemia
* History of arterial thrombotic events (myocardial infarction, stroke or peripheral vascular disease).
* Uncontrolled hypertension
* Taking medications that are known to be associated with Torsades de Pointes
* Ongoing active infection
* Diagnosed with or received anti-cancer therapy for another primary malignancy within 3 years prior to entry (except for non-melanoma skin cancer or in situ cancers)
* Any condition or illness tha could compromise patient safety or interfere with the evaluation of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, Irvine, Orange, California
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Wu H, Shih JY, Yang JC. Rapid Response to Sunitinib in a Patient with Lung Adenocarcinoma Harboring KIF5B-RET Fusion Gene. J Thorac Oncol. 2015 Sep;10(9):e95-e96. doi: 10.1097/JTO.0000000000000611. No abstract available. PMID 26291023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ponatinib Treatment Arm
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 58 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Asian | 0
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The number of participants that achieved either a partial or complete response assessed using Response Evaluation Criteria in Solid Tumors (RECIST v 1.1)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the start of treatment until disease progression or death, up to approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Disease Control Rate
Description: The number of participants that achieved either a partial or complete response or stable disease, assessed using Response Evaluation Criteria in Solid Tumors (RECIST v 1.1)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: From the start of treatment until disease progression or death, up to approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Participants | 5

3. Secondary Outcome: Median Progression-Free Survival
Description: The duration of time from study entry until disease progression (assessed using RECIST 1.1.) or death.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression.
Time Frame: From study entry until disease progression or death, median duration of 3.8 months
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Months | 3.8 [1.83 to 5.3]

4. Secondary Outcome: 1 Year Overall Survival Rate
Description: The number of participants surviving one year after study entry
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Participants | 5

5. Secondary Outcome: Number of Participants With Adverse Events
Description: The number of participants with grade 3 plus adverse events as assessed using Common Toxicology Criteria for Adverse Events (CTCAE 4) that were deemed to be possibly, probably, or definitely related to study treatment.
Time Frame: From the start of treatment until 30 days after the end of treatment (up to approximately 2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Ponatinib Treatment Arm
Number analyzed (Participants) | 9
Participants | 2

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment (up to approximately 2 years)
Arm/Group | Ponatinib Treatment Arm
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib Treatment Arm (N=9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib Treatment Arm (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (6)
Pain (General disorders) | 4 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (7)
Hypothyroidism (Endocrine disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (4)
Bronchial infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2)
Blurred vision (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT01813734/Prot_SAP_000.pdf